CLINICAL TRIAL: NCT05873309
Title: The Role of OXytocin in Acute Ischemic Stroke reconvAlesceNcE: The ROXANE Study
Acronym: ROXANE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Academy of Medical Sciences (SAMS) (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00608; ko23katan
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
Keywords: oxytocin; blood biomarkers
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evidence suggests that oxytocin has a neuroprotective role on a systemic and cellular level in the context of acute ischemic stroke (AIS). The investigators therefore hypothesize that high levels of circulating oxytocin measured within the first 72 hours after symptom onset are associated with lower mortality and favorable outcome in acute ischemic stroke.

DETAILED DESCRIPTION:
The preliminary data suggest a possible neuroprotective role of oxytocin via endocrine as well as paracrine effects, underscoring that oxytocin levels in the acute phase of stroke may have a considerable influence on patient outcomes. However, the role of oxytocin in acute ischemic stroke patients has, to our knowledge, never been investigated. If oxytocin really shows a strong associated with functional outcomes after stroke and given the fact that commercially available oxytocin can be safely administered via nasal spray, oxytocin would become an innovative and highly interesting novel therapeutic agent for ischemic stroke patients in the near future. For the ROXANE cohort the investigators plan to recruit patients with acute ischemic stroke from the University Hospital in Basel. The study is designed as an observational cohort study, because an observational study is currently at this stage of knowledge (effect of oxytocin in vitro and in vivo (animal models)), the best study design. It harbors minimal harm, but still allows us to adequately estimate the association of oxytocin levels in humans with stroke outcome. If it is possible to establish this association in humans based on results of the planned observation study, the investigators will be able to plan an interventional trial, which may directly beneficially impact clinical outcome of stroke patient.

ELIGIBILITY:
Inclusion Criteria:

* Rapid onset of a focal neurologic deficit, with signs or symptoms persisting beyond 24 hours and not associated with infection, trauma, or tumor of the brain, severe metabolic disorders, or chronic degenerative neurologic disease; or
* the development of an acute focal neurologic deficit persisting >24 hours in conjunction with brain imaging consistent with acute ischemic stroke. The CT or MRI may either show a new infarct or no change from the study performed at entry, i.e., the diagnosis is clinical and does not require CT/MRI confirmation. Secondary hemorrhagic infarction is permissible.
* First blood sample at the stroke unit is taken within 24 hours from symptom onset.

Exclusion Criteria:

* Patients below 18 years
* Hemorrhagic stroke or patients discharged from the hospital with a diagnosis different from ischemic stroke (i.e., stroke mimics)
* Missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the ROXANE cohort the investigators plan to recruit patients with acute ischemic stroke from the University Hospital in Basel.
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
90-day mortality Rate | 90 days after stroke
  The 90-day mortality rate will be assessed via a structured telephone interview on day 90 (+/- 10)
90-day functional outcome | 90 days after stroke
  The 90-day functional outcome will be assessed with the modified Ranking Scale (mRS) via a structured telephone interview on day 90 (+/- 10). The modified Ranking Scale is a 6 point disability scale with possible scores ranging from 0 to 5. 0= no symptoms, 5 = severe disability. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. A favorable outcome is defined as a mRS score of 0 to 2 points.

SECONDARY OUTCOMES:
Assessment of post-stroke symptoms | 90 days after stroke
  Patient Health Questionnaire-9 (PHQ-9) will be assessed via a structured telephone interview. The PHQ-9 is scored 0 to 27, with scores >/= 10 indicating a possible depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Frenger, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No